CLINICAL TRIAL: NCT02437240
Title: Effects of Pilates-based Cardiopulmonary Physical Therapy for In-Patients After Cardiac Surgery
Brief Title: Pilates-based Cardiopulmonary Physical Therapy for In-Patients After Cardiac Surgery
Acronym: PBCPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Mei-Wun Tsai, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NationalYangMingU
Record Dates: First submitted 2015-04-16; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Other Functional Disturbances Following Cardiac Surgery
Keywords: Pilates-based exercise; respiratory mechanics; cardiopulmonary physical therapy; sternotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilates-based CPT (Experimental): incorporated the concept of pilates training into cardiopulmonary physical therapy after cardiac surgery
  Interventions: Behavioral: Pilates-based CPT
- Traditional CPT (Active Comparator): usual bed side cardiopulmonary physical therapy after cardiac surgery
  Interventions: Behavioral: Traditional CPT

INTERVENTIONS:
Behavioral: Pilates-based CPT — To emphasize the self-perception of breathing and body core control during in-patient cardiopulmonary physical therapy following cardiac surgery
  Arms: Pilates-based CPT
Behavioral: Traditional CPT — A traditional in-patient cardiopulmonary physical therapy following cardiac surgery including airway clearance, breathing exercises, chest mobility and reconditioning exercises and so on
  Arms: Traditional CPT

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of pilates-based cardiopulmonary physical therapy (CPT) for in-patients after cardiac surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary and musculoskeletal complications are the most frequent and significant contributor to morbidity, mortality with hospitalization. Pilates-based exercise has be applied to improve core control, movement efficiency and postural stability. High incidence of musculoskeletal problems have been concerned in relation to the patient's functional recovery after cardiac surgery. However, no literature is addressed how to manage this issue effectively till now. The purpose of this clinical trial is to evaluate the effect of pilates-based cardiopulmonary physical therapy for in-patients after cardiac surgery. This is a single-blinded, randomized control trial. Investigators will enroll pre-cardiac surgery and allocate subjects to modified Pilates-based training group or control group using block randomization.The training protocol will be based on pilates concepts. The control group is treated with a conventional protocol of physical therapy. The study will be carried on whole in-patient phase. During this period, patients received respiratory motion analysis, chest wall muscles mobility, lung function and endurance evaluation. Patients' changes in respiratory movement, cardiopulmonary endurance, and lung function will be evaluated by an assessor blinded to the intervention at admission and discharge from hospital. After 6 months after hospital discharge, patient's respiratory motion, lung function and disease specific health related quality of life will be evaluated. All outcomes will be described by mean (SD) or number (%). Independent t test or chi square test will be used to compare the basic data difference between training group and conventional group. Then, two-way analysis of variance or two-way analysis of covariance will be used to compare the outcomes difference between groups. Alpha level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* post open heart surgery
* FVC> 80% of predicted and/or FEV1>70% of predicted
* age >/=20 years old
* approve inform consent

Exclusion Criteria:

* preoperative severe pulmonary hypertension
* moderate to severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease
* heart failure or s/p heart transplant
* emergent surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
change from pre-operation in respiratory mechanics | at hospital discharge, an expected average of 2 weeks after surgery
  Chest motion in deep breathing will be assessed simultaneously by 3D reality motion analysis and spirometer. Participants will be followed at hospital discharge, an expected average of 2 weeks after surgery.

SECONDARY OUTCOMES:
change from pre-operation in respiratory mechanics | at 6 month after surgery
  Chest motion in deep breathing will be assessed simultaneously by 3D reality motion analysis and spirometer. Participants will be followed at 6 month after surgery.
change from pre-operation in chest mobility | at hospital discharge, an expected average of 2 weeks after surgery
  Chest mobility will be assessed by tape measuring the difference of chest circumference between deep inspiration and expiration. Participants will be followed at hospital discharge, an expected average of 2 weeks after surgery.
abnormal breathing pattern | at hospital discharge, an expected average of 2 weeks after surgery
  Abnormal breathing pattern will be assessed by physical examination and camera recording if there is any paradoxical, asymmetrical chest movements during breathing. Participants will be followed at hospital discharge, an expected average of 2 weeks after surgery.
abnormal breathing pattern | at 6 month after surgery
  Abnormal breathing pattern will be assessed by physical examination and camera recording if there is any paradoxical, asymmetrical chest movements during breathing. Participants will be followed at 6 month after surgery.
Percentage change from preoperative pulmonary function | at hospital discharge, an expected average of 2 weeks after surgery
  Percentage of preoperative pulmonary function, including forced vital capacity (FVC), the first second forced expiratory volume (FEV1), peak inspiratory flow and peak expiratory flow are measured by spirometry at hospital discharge, an expected average of 2 weeks after cardiac surgery
Percentage change from preoperative pulmonary function | at 6 month after surgery
  Percentage of preoperative pulmonary function, including forced vital capacity (FVC), the first second forced expiratory volume (FEV1), peak inspiratory flow and peak expiratory flow are measured by spirometry at 6 month after surgery
change of cardiopulmonary fitness | at hospital discharge, an expected average of 2 weeks after cardiac surgery
  Six-minute walking test is used to assess cardiopulmonary fitness at hospital discharge, an expected average of 2 weeks after cardiac surgery.
cardiopulmonary exercise function | at one month after hospital discharge
  Symptom-limited graded exercise testing is used to assess cardiopulmonary exercise function at one month after hospital discharge.
health related quality of life | at 6 month after hospital discharge
  Cardiovascular Limitations and Symptoms Profile (37 items) is used to assess disease specific health related quality of life at 6 month after hospital discharge.

REFERENCES:
- [Background] Grover FL, Cleveland JC Jr, Shroyer LW. Quality improvement in cardiac care. Arch Surg. 2002 Jan;137(1):28-36. doi: 10.1001/archsurg.137.1.28. PMID 11772211
- [Background] Lunardi AC, Marques da Silva CC, Rodrigues Mendes FA, Marques AP, Stelmach R, Fernandes Carvalho CR. Musculoskeletal dysfunction and pain in adults with asthma. J Asthma. 2011 Feb;48(1):105-10. doi: 10.3109/02770903.2010.520229. Epub 2010 Dec 29. PMID 21189115
- [Background] Kantor E, Poupard L, Le Bozec S, Bouisset S. Does body stability depend on postural chain mobility or stability area? Neurosci Lett. 2001 Aug 3;308(2):128-32. doi: 10.1016/s0304-3940(01)01986-3. PMID 11457576
- [Background] Perri M. Pain and Faulty Breathing: A Pilot Study. J Bodywork & Mov Ther. 2004 (8): 297-306.
- [Background] Sasseron AB, Figueiredo LC, Trova K, Cardoso AL, Lima NM, Olmos SC, Petrucci O. Does the pain disturb the respiratory function after open heart surgery? Rev Bras Cir Cardiovasc. 2009 Oct-Dec;24(4):490-6. doi: 10.1590/s0102-76382009000500010. English, Portuguese. PMID 20305922
- [Background] Wynne R, Botti M. Postoperative pulmonary dysfunction in adults after cardiac surgery with cardiopulmonary bypass: clinical significance and implications for practice. Am J Crit Care. 2004 Sep;13(5):384-93. PMID 15470854
- [Background] Basoglu OK, Atasever A, Bacakoglu F. The efficacy of incentive spirometry in patients with COPD. Respirology. 2005 Jun;10(3):349-53. doi: 10.1111/j.1440-1843.2005.00716.x. PMID 15955148
- [Background] Gosselink R, Schrever K, Cops P, Witvrouwen H, De Leyn P, Troosters T, Lerut A, Deneffe G, Decramer M. Incentive spirometry does not enhance recovery after thoracic surgery. Crit Care Med. 2000 Mar;28(3):679-83. doi: 10.1097/00003246-200003000-00013. PMID 10752814
- [Background] Carvalho CR, Paisani DM, Lunardi AC. Incentive spirometry in major surgeries: a systematic review. Rev Bras Fisioter. 2011 Sep-Oct;15(5):343-50. doi: 10.1590/s1413-35552011005000025. Epub 2011 Oct 14. PMID 22002191
- [Background] Pilates JH 1988 Your Health. Revised edition. Robbins J (ed). Presentation Dynamics, Incline Village, NV. First published, 1934
- [Background] Rogers K, Gibson AL. Eight-week traditional mat Pilates training-program effects on adult fitness characteristics. Res Q Exerc Sport. 2009 Sep;80(3):569-74. doi: 10.1080/02701367.2009.10599595. PMID 19791643
- [Background] Segal NA, Hein J, Basford JR. The effects of Pilates training on flexibility and body composition: an observational study. Arch Phys Med Rehabil. 2004 Dec;85(12):1977-81. doi: 10.1016/j.apmr.2004.01.036. PMID 15605336
- [Background] Sorosky S, Stilp S, Akuthota V. Yoga and pilates in the management of low back pain. Curr Rev Musculoskelet Med. 2008 Mar;1(1):39-47. doi: 10.1007/s12178-007-9004-1. PMID 19468897
- [Background] Herrington L, DaviesR. The influence of Pilates training on the ability to contract the Transversus Abdominis muscle in asymptomatic individuals. J Bodyw Mov Ther 2005;9:52-7
- [Background] Culligan PJ, Scherer J, Dyer K, Priestley JL, Guingon-White G, Delvecchio D, Vangeli M. A randomized clinical trial comparing pelvic floor muscle training to a Pilates exercise program for improving pelvic muscle strength. Int Urogynecol J. 2010 Apr;21(4):401-8. doi: 10.1007/s00192-009-1046-z. Epub 2010 Jan 22. PMID 20094704
- [Background] Cruz-Ferreira A, Fernandes J, Laranjo L, Bernardo LM, Silva A. A systematic review of the effects of pilates method of exercise in healthy people. Arch Phys Med Rehabil. 2011 Dec;92(12):2071-81. doi: 10.1016/j.apmr.2011.06.018. Epub 2011 Oct 24. PMID 22030232
- [Background] Johnson EG, Larsen A, Ozawa H, Wilson CA, Kennedy KL. The effects of Pilates-based exercise on dynamic balance in healthy adults. J Bodyw Mov Ther 2007;11:238-42
- [Background] Irez GB, Ozdemir RA, Evin R, Irez SG, Korkusuz F. Integrating pilates exercise into an exercise program for 65+ year-old women to reduce falls. J Sports Sci Med. 2011 Mar 1;10(1):105-11. eCollection 2011. PMID 24149302
- [Background] Endleman I, Critchley DJ. Transversus abdominis and obliquus internus activity during pilates exercises: measurement with ultrasound scanning. Arch Phys Med Rehabil. 2008 Nov;89(11):2205-12. doi: 10.1016/j.apmr.2008.04.025. PMID 18996251
- [Background] Emery K, De Serres SJ, McMillan A, Cote JN. The effects of a Pilates training program on arm-trunk posture and movement. Clin Biomech (Bristol). 2010 Feb;25(2):124-30. doi: 10.1016/j.clinbiomech.2009.10.003. Epub 2009 Oct 30. PMID 19879677
- [Background] Queiroz BC, Cagliari MF, Amorim CF, Sacco IC. Muscle activation during four Pilates core stability exercises in quadruped position. Arch Phys Med Rehabil. 2010 Jan;91(1):86-92. doi: 10.1016/j.apmr.2009.09.016. PMID 20103401
- [Background] Brooks-Brunn JA. Postoperative atelectasis and pneumonia: risk factors. Am J Crit Care. 1995 Sep;4(5):340-9; quiz 350-1. PMID 7489036
- [Background] Hirschhorn AD, Richards D, Mungovan SF, Morris NR, Adams L. Supervised moderate intensity exercise improves distance walked at hospital discharge following coronary artery bypass graft surgery--a randomised controlled trial. Heart Lung Circ. 2008 Apr;17(2):129-38. doi: 10.1016/j.hlc.2007.09.004. Epub 2007 Dec 3. PMID 18060837
- [Background] Stein R, Maia CP, Silveira AD, Chiappa GR, Myers J, Ribeiro JP. Inspiratory muscle strength as a determinant of functional capacity early after coronary artery bypass graft surgery. Arch Phys Med Rehabil. 2009 Oct;90(10):1685-91. doi: 10.1016/j.apmr.2009.05.010. PMID 19801057
- [Background] Hedenstierna G, Edmark L. Mechanisms of atelectasis in the perioperative period. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):157-69. doi: 10.1016/j.bpa.2009.12.002. PMID 20608554
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Hodges PW, Gurfinkel VS, Brumagne S, Smith TC, Cordo PC. Coexistence of stability and mobility in postural control: evidence from postural compensation for respiration. Exp Brain Res. 2002 Jun;144(3):293-302. doi: 10.1007/s00221-002-1040-x. Epub 2002 Apr 13. PMID 12021811
- [Background] CH Hsu, YC Chung, LY Kuo, JC Chen, FH Chen, HY Huang. Respiratory effects on cardiac rehabilitation combined Pilates exercise in patients underwent cardiac surgery. Formosan Journal of Physical Therapy 2013; 38(3): 210-218
- [Result] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 1--coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S2-22. doi: 10.1016/j.athoracsur.2009.05.053. PMID 19559822
- See also: Postoperative complications among patients undergoing cardiac surgery — http://WWW.UPTODATE.COM